CLINICAL TRIAL: NCT02142920
Title: A Phase One, Open-Label Single-Radiolabeled Dose Study To Investigate The Metabolism, And Excretion Of [14c]-PF-05212384 In Healthy Male Volunteers
Brief Title: Investigation Of The Metabolism, And Excretion Of [14c]-PF-05212384 In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2151006
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C] PF 05212384 (Experimental): Receive PF-05212384 89 mg Dose
  Interventions: Drug: PF-05212384

INTERVENTIONS:
Drug: PF-05212384 — Single 89 mg Dose via 30 minute IV infusion

SUMMARY:
The purpose of the study is to characterize how PF-05212384 is metabolized in the body following a single intravenous dose of radioactively labeled drug ([14C]-PF-05212384).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 30- 65 years vasectomised or >40 with no desire to father children in the near future (12 months), inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects agree to use an adequate method of contraception

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen or history of drug or alcohol abuse in the past 2 years.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0.5 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0.5 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 9 Days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area under the Concentration-Time Curve (AUC) | 9 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Plasma Decay Half-Life (t1/2) | 9 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Systemic Clearance (CL) | 9 days
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution at Steady State (Vss) | 9 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ruddington Fields, Nottingham, United Kingdom

REFERENCES:
- [Derived] Houk BE, Alvey CW, Visswanathan R, Kirkovsky L, Matschke KT, Kimoto E, Ryder T, Obach RS, Durairaj C. Distribution, Metabolism, and Excretion of Gedatolisib in Healthy Male Volunteers After a Single Intravenous Infusion. Clin Pharmacol Drug Dev. 2019 Jan;8(1):22-31. doi: 10.1002/cpdd.615. Epub 2018 Sep 26. PMID 30256541
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2151006&StudyName=Investigation%20Of%20The%20Metabolism%2C%20And%20Excretion%20Of%20%5B14c%5D-PF-05212384%20In%20Healthy%20Male%20Volunteers%20